CLINICAL TRIAL: NCT01971606
Title: Impact of High-dose Pretreatment of Rosuvastatin in Patients With Acute Coronary Syndrome Following Off-pump Coronary Artery Bypass: Results From the HIROP-ACS (HIgh-dose Pretreatment of Rosuvastatin During Off-Pump Coronary Bypass in Acute Coronary Syndrome) Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 4-2007-0253
Record Dates: First submitted 2013-10-23; First posted 2013-10-29 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: A Total of 234 Patients With Acute Coronary Syndrome Who Will Undergo OPCAB.
Keywords: Statin, coronary artery bypass grafting, off-pump surgery, acute coronary syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rosuvastatin group (Experimental): Rosuvastatin group
  Interventions: Drug: Rosuvastatin
- Placebo group (Placebo Comparator): Placebo group
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin — Patients will be randomized in a ratio of 1:1 to A) High-dose rosuvastatin vs. B) Placebo.
  A) Rosuvastatin group : Administration of 40mg of rosuvastatin PO 12 hours before surgery and 20mg of rosuvastatin PO 2hours before surgery and 10mg of rosuvastatin PO daily at postoperative period.
  B) Placebo group : Administration of placebo at 12 hours and 2 hours before surgery and 10mg of rosuvastatin PO daily at postoperative period.

SUMMARY:
Periprocedural treatment with high-dose statins is known to have cardioprotective and pleiotropic effects, such as anti-thrombotic and anti-inflammatory actions.

-Objective: to determine whether preoperative rosuvastatin loading is independently associated with reduced myocardial ischemia and clinical outcomes in patients with stable angina undergoing isolated off-pump coronary bypass (OPCAB) in patients with acute coronary syndrome.

Study design

* Prospective, double-blinded, single-center study of each 117 subjects enrolled
* Subjects with acute coronary syndrome who meet all inclusion and exclusion criteria will be enrolled preoperatively.
* Eligible subjects will be randomized 1:1 to A) High-dose rosuvastatin (n=117) vs. B) Placebo (n=117).
* The amount of preoperative administration of high-dose rosuvastatin will be 60mg of a total
* All subjects will undergo OPCAB procedure. - The primary and secondary endpoints will be compared at 30 days and 2 years postoperatively between two groups

ELIGIBILITY:
Inclusion Criteria:

* The presence of acute coronary syndrome, including unstable angina, acute non-ST elevation myocardial infarction
* Age of 19 years or older
* A need for isolated surgical myocardial revascularization
* Patients with signed informed consent

Exclusion Criteria:

* Patients with combined surgery with coronary bypass grafting
* On-pump conversion
* Patients with any increase in liver enzymes
* Patients with history of liver or muscle disease.
* Patients with moderate renal dysfunction (creatinine>2.0mg/dl) or need for dialysis
* Re-do surgery
* Urgent/emergent surgery

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2007-10; Primary Completion 2012-06 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac events (MACEs) | 30 days after OPCAB
  Major adverse cardiac events (MACEs), which include the following: death from all causes, non-fatal myocardial infarction (MI), and repeat revascularization by percutaneous intervention or bypass surgery within 30 days after OPCAB.

SECONDARY OUTCOMES:
The degree of myocardial ischemia and inflammatory | immediate, 24 hours, 48 hours, 72 hours, 7 days after OPCAB
  The degree of myocardial ischemia and inflammatory changes assessed by blood sampling and specific tests (CK-MB, Troponin T, ESR, CRP, hs-CRP) at the early period after OPCAB.

OTHER OUTCOMES:
Incidence of postoperative atrial arrhythmia including atrial fibrillation and atrial flutter | 30 days after OPCAB
Incidence of postoperative renal impairment or a need for dialysis | 30 days after OPCAB
Late MACEs 2 years after OPCAB | 2 years after OPCAB

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiovascular Surgery, Severance Cardiovascular Hospital , Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Background] Patti G, Pasceri V, Colonna G, Miglionico M, Fischetti D, Sardella G, Montinaro A, Di Sciascio G. Atorvastatin pretreatment improves outcomes in patients with acute coronary syndromes undergoing early percutaneous coronary intervention: results of the ARMYDA-ACS randomized trial. J Am Coll Cardiol. 2007 Mar 27;49(12):1272-8. doi: 10.1016/j.jacc.2007.02.025. PMID 17394957